CLINICAL TRIAL: NCT00161161
Title: Genetic Liability in the Brain Morphology of Attention Deficit Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: The Dutch Brain Foundation (Other)
Other Study IDs: WOM 99/076
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-12-30 (Estimated); Status verified 2005-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; MRI; genetics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a heritable psychiatric disorder with onset in childhood. Twin and adoption studies indicate that additive genetic factors explain up to 80% of the variance underlying susceptibility. The siblings of children with ADHD have a three- to fivefold increased risk of having ADHD compared to the siblings of healthy control subjects, and the risk is even greater for monozygotic twins with 50-80% concordance compared with up to 33% in dizygotic twins). As full siblings share on average 50% of their genes, even the unaffected siblings of children with ADHD would be expected to share some of the genes involved in the disorder. The neuroanatomical substrate of ADHD is becoming increasingly better defined by a growing body of evidence from imaging studies. Evidence from neuroimaging studies suggests that this disorder is associated with reductions in brain volume up to 5% in these children. In this protocol we collected MRI-scans from boys with ADHD and their unaffected siblings, as well as control subjects. In addition, cheekswabs were later collected for DNA analysis.

ELIGIBILITY:
Inclusion Criteria:

1. age 7 - 18 years.

Inclusion criteria for patients

1. DSM-IV (APA, 1994) diagnosis of ADHD (combined subtype), according to DISC interview
2. scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form (TRF)
3. one brother who meets the inclusion criteria for siblings

Inclusion criteria for siblings

1. no DSM-IV (APA,1994) diagnosis for ADHD or another disruptive disorder (ODD or CD), according to DISC interview
2. no scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form (TRF)

Inclusion criteria for controls

1. no DSM-IV (APA, 1994) diagnosis, according to DISC interview
2. no scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form (TRF)

Exclusion Criteria:

1. IQ < 70
2. illness of the cardiovascular, the endocrine, the pulmonal or the gastrointestinal system
3. the presence of metal objects in or around the body (pacemaker, dental braces)

Ages: 7 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90
Dates: Start 1999-10; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Durston, Ph.D., Principal Investigator — RMI of Neuroscience, UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Durston S, Hulshoff Pol HE, Schnack HG, Buitelaar JK, Steenhuis MP, Minderaa RB, Kahn RS, van Engeland H. Magnetic resonance imaging of boys with attention-deficit/hyperactivity disorder and their unaffected siblings. J Am Acad Child Adolesc Psychiatry. 2004 Mar;43(3):332-40. doi: 10.1097/00004583-200403000-00016. PMID 15076267
- [Result] Durston S, Fossella JA, Casey BJ, Hulshoff Pol HE, Galvan A, Schnack HG, Steenhuis MP, Minderaa RB, Buitelaar JK, Kahn RS, van Engeland H. Differential effects of DRD4 and DAT1 genotype on fronto-striatal gray matter volumes in a sample of subjects with attention deficit hyperactivity disorder, their unaffected siblings, and controls. Mol Psychiatry. 2005 Jul;10(7):678-85. doi: 10.1038/sj.mp.4001649. PMID 15724142